CLINICAL TRIAL: NCT01854125
Title: Efficacy of Autologous Mesenchymal Stem Cell Transplantation Via Liver Artery in Liver Cirrhosis Patients With Refractory Ascites
Brief Title: Autologous Mesenchymal Stem Cell Transplantation in Cirrhosis Patients With Refractory Ascites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shihui, Department of Gastroenterology and Hepatology, Nanjing PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NanjingPLAGH1; Jinling 01 (Other: Jinling Hospital)
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Immune Function in Blood; Liver Function in Blood; Variation of Ascites; Characters of Quality of Life; Child-Pugh Score
Keywords: immun function; liver function; ascites; quality of life; Child-Pugh score
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- autologous bone marrow mesenchymal stem cells transplantation (Active Comparator): Every patient is given 1x106 MSCs per kg infused via liver artery
  Interventions: Biological: autologous bone marrow mesenchymal stem cells transplantation; Biological: autologous bone marrow msenchymal stem cells transplantation
- mesenchymal stem cells transplantation (Active Comparator): autologous bone marrow mesenchymal stem cells transplantation
  Interventions: Biological: autologous bone marrow mesenchymal stem cells transplantation; Biological: autologous bone marrow msenchymal stem cells transplantation
- stem cells transplantation (Experimental): autologous bone marrow mesenchymal stem cells transplantation
  Interventions: Biological: autologous bone marrow mesenchymal stem cells transplantation; Biological: autologous bone marrow msenchymal stem cells transplantation

INTERVENTIONS:
Biological: autologous bone marrow mesenchymal stem cells transplantation — Autologous MSCs were infused to patients using interventional method via hepatic artery . The catheter was inserted to proper hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography, autologous bone marrow MSCs were infused slowly for 20-30 minutes.
Biological: autologous bone marrow msenchymal stem cells transplantation

SUMMARY:
Liver cirrhosis (LC) is the final destiny in chronic liver disease.The quality of life in liver cirrhosis patients with refractory ascites are very wretched. The objective of this study is to evaluate the therapeutic efficacy of autologous bone marrow mesenchymal stem cells (BMSCs) transplantation via liver artery in Child-Pugh B and C stage of liver cirrhosis patients with refractory ascites. The immunomodulatory impact of MSCs in fibrosis was confirmed, and several clinical studies have applied MSCs to eliminate the progression of fibrosis. In this research the investigators will study the affect and influence of MSCs in the patients,include assay of liver function,variation of ascites,Child-Pugh score etc.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

Aged 18~65 years. Ultrasonographic evidences of cirrhosis. hepatic cirrhosis patients with refractory ascite.

Exclusion Criteria:

history of moderate to severe hepatic encephalopathy or variceal bleeding during the last two months before enrolment.

Prothrombin time is less than 30s. Severe problems in other vital organs(e.g.the heart,renal or lungs). Liver tumor on ultrasonography, CT or MRI examination. Pregnant or lactating women. Imaging evidences of vascular thromboses.

-

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
change in immune function,liver function in blood | before and one to 12 weeks after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Fangyu Wang, MD/PhD, Study Director — Nanjing University; Fangyu Wang, MD/PhD, Study Director — Nanjin University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Kharaziha P, Hellstrom PM, Noorinayer B, Farzaneh F, Aghajani K, Jafari F, Telkabadi M, Atashi A, Honardoost M, Zali MR, Soleimani M. Improvement of liver function in liver cirrhosis patients after autologous mesenchymal stem cell injection: a phase I-II clinical trial. Eur J Gastroenterol Hepatol. 2009 Oct;21(10):1199-205. doi: 10.1097/MEG.0b013e32832a1f6c. PMID 19455046